CLINICAL TRIAL: NCT02195375
Title: A Randomised Double-blind, Double-dummy Parallel Group Study to Compare the Efficacy and Safety of Fluticasone Propionate / Formoterol Fumarate (Flutiform®) 500/20 µg BID and 250/10 µg BID Versus Salmeterol / Fluticasone (Seretide®) 50/500 µg BID in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Flutiform® Compared With Seretide® in the Treatment of COPD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLT3510
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; FEV1 ≤ 50%
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone-formoterol; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Flutiform 500/20 µg BID (Experimental): Flutiform 250/10 (2 puffs BID)
  Interventions: Drug: Flutiform 500/20 µg BID
- Flutiform 250/10 µg BID (Experimental): Flutiform 125/5 (2 puffs BID)
  Interventions: Drug: Flutiform 250/10 µg BID
- Seretide Accuhaler 50/500 µg BID (Active Comparator): Seretide Accuhaler 50/500 (BID)
  Interventions: Drug: Seretide Accuhaler 50/500 µg BID

INTERVENTIONS:
Drug: Flutiform 500/20 µg BID
  Arms: Flutiform 500/20 µg BID
Drug: Flutiform 250/10 µg BID
  Arms: Flutiform 250/10 µg BID
Drug: Seretide Accuhaler 50/500 µg BID
  Arms: Seretide Accuhaler 50/500 µg BID

SUMMARY:
The purpose of this study is to investigate whether flutiform® is effective and safe in the treatment of chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
A multi-centre, randomised, double-blind, double dummy, active-controlled, parallel-group study in male and female subjects conducted to assess the efficacy and safety of flutiform in the treatment of COPD. Subjects will be randomised to one of three treatment groups in a 1:1:1 ratio. Throughout the study subjects will be assessed on a mixture of symptom based and lung function measurements to monitor their progress in the study.

ELIGIBILITY:
Inclusion:

1. Male or Female subjects aged ≥ 40 years at screening visit.
2. Diagnosis of COPD
3. Willing and able to replace current COPD therapy with study medication.
4. Able to demonstrate correct use of a pMDI with or without a spacer and Accuhaler.
5. Willing and able to attend all study visits and complete study assessments.
6. Able to provide signed informed consent.

Exclusion:

1. Ongoing moderate or severe exacerbation of COPD in the 2 weeks before screening.
2. Current diagnosis of asthma.
3. Documented evidence of α1-antitrypsin deficiency as the underlying cause of COPD.
4. Other active respiratory disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung disease, cystic fibrosis, bronchiolitis obliterans.
5. Previous lung resection.
6. Use of long-term oxygen therapy (LTOT) or mechanical ventilation. Note: LTOT is defined as >15 hours use per day
7. Chest X-ray or CT scan that reveals evidence of clinically significant abnormalities not believed to be due to COPD.
8. Evidence of uncontrolled cardiovascular disease.
9. Evidence of clinically significant renal, hepatic, gastrointestinal, or psychiatric disease.
10. Current malignancy or a previous history of cancer which has been in remission for < 5 years (basal cell or squamous cell carcinoma of the skin which has been resected is not excluded).
11. Clinically significant sleep apnoea requiring use of continuous positive airway pressure (CPAP) device or non-invasive positive pressure ventilation (NIPPV) device.
12. Participation in the acute phase of a pulmonary rehabilitation programme within 4 weeks prior to screening or during the study.
13. Known or suspected history of drug or alcohol abuse in the last 2 years.
14. Requiring treatment with any of the prohibited concomitant medications.
15. Known or suspected hypersensitivity to study drug or excipients.
16. Received an investigational drug within 30 days of the screening visit (12 weeks if an oral or injectable steroid).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 923 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Average pre-dose FEV1 | 26 weeks

SECONDARY OUTCOMES:
Average 1 hour Post dose FEV1, FVC, FEV6 | 26 Weeks

OTHER OUTCOMES:
Moderate and Severe COPD Exacerbations | 26 weeks
COPD Assessment Test | Change from baseline to week 8, week 14, week 26
Average capacity of daily living during the morning score | 26 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Fitzroy, Australia
- Beijing, China
- Wellington, New Zealand
- Seoul, South Korea
- Taipei, Taiwan